CLINICAL TRIAL: NCT04819958
Title: The Effect of Immunological Heterogeneity of Tumor Microenvironment in the Short-term Outcome and Long-term Outcome of Patients With Gastric Cancer
Brief Title: The Effect of Immunological Heterogeneity of Tumor Microenvironment in the Prognosis of Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Head of Department of Gastric Surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Other Study IDs: FUGES-B01
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the resected specimens with DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to explore the effect of immunological heterogeneity of tumor microenvironment in the short-term outcome and long-term outcome of patients with gastric cancer.

DETAILED DESCRIPTION:
A prospective cohort study will be performed to explore the effect of immunological heterogeneity of tumor microenvironment in the short-term outcome and long-term outcome of patients with gastric cancer. The evaluation parameters are perioperative clinical efficacy, postoperative complications, and 3-year survival and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 80 years
2. Histology confirmed gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy.
3. Clinical stage: cTNM: stage I or above at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Eighth Edition
4. Performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 2 (normal to symptomatic but in bed less than half the day)
5. Clinically fit for gastric cancer surgery, i.e. adequate renal, hepatic, hematologic, and pulmonary function.
6. Written informed consent

Exclusion Criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of previous gastrectomy, endoscopic mucosal resection, or endoscopic submucosal dissection
4. History of other malignant diseases within the past five years
5. History of unstable angina or myocardial infarction within the past six months
6. History of a cerebrovascular accident within the past six months
7. History of continuous systematic administration of corticosteroids within one month
8. Requirement of simultaneous surgery for other diseases
9. Emergency surgery due to complication (bleeding, obstruction, or perforation) caused by gastric cancer
10. Forced expiratory volume in 1 second (FEV1)<50% of predicted values
11. Inclusion in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are assigned to undergo gastrectomy for gastric cancer are included.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months
  3-year disease free survival rate

SECONDARY OUTCOMES:
3-year overall survival rate | 36 months
  3-year overall survival rate
Morbidity rates | 30 days
  This is for the incidence of early postoperative complications, which defined as the event observed within 30 days after surgery.
Mortality rates | 30 days
  This is for the early mortality, which defined as the event observed within 30 days after surgery.
Total number of retrieved lymph nodes | One month after surgery
  Total number of retrieved lymph nodes after surgery
Intraoperative morbidity rates | 1 day
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
The variation of white blood cell count | Preoperative 7 days and postoperative 1, 3, and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of hemoglobin | Preoperative 7 days and postoperative 1, 3, and 5 days
  The values of hemoglobin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of C-reactive protein | Preoperative 7 days and postoperative 1, 3, and 5 days
  The values of C-reactive protein in milligram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into four categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, and mixed type
Time to first ambulation | 30 days
  Time to first ambulation in days is used to assess the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus in days is used to assess the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet in days is used to assess the postoperative recovery course.
Time to first soft diet | 30 days
  Time to first soft diet in days is used to assess the postoperative recovery course.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastric Surgery, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumagai S, Togashi Y, Kamada T, Sugiyama E, Nishinakamura H, Takeuchi Y, Vitaly K, Itahashi K, Maeda Y, Matsui S, Shibahara T, Yamashita Y, Irie T, Tsuge A, Fukuoka S, Kawazoe A, Udagawa H, Kirita K, Aokage K, Ishii G, Kuwata T, Nakama K, Kawazu M, Ueno T, Yamazaki N, Goto K, Tsuboi M, Mano H, Doi T, Shitara K, Nishikawa H. The PD-1 expression balance between effector and regulatory T cells predicts the clinical efficacy of PD-1 blockade therapies. Nat Immunol. 2020 Nov;21(11):1346-1358. doi: 10.1038/s41590-020-0769-3. Epub 2020 Aug 31. PMID 32868929
- [Background] Smyth EC, Nilsson M, Grabsch HI, van Grieken NC, Lordick F. Gastric cancer. Lancet. 2020 Aug 29;396(10251):635-648. doi: 10.1016/S0140-6736(20)31288-5. PMID 32861308
- [Background] Utzschneider DT, Gabriel SS, Chisanga D, Gloury R, Gubser PM, Vasanthakumar A, Shi W, Kallies A. Early precursor T cells establish and propagate T cell exhaustion in chronic infection. Nat Immunol. 2020 Oct;21(10):1256-1266. doi: 10.1038/s41590-020-0760-z. Epub 2020 Aug 24. PMID 32839610
- [Background] Gao Y, Nihira NT, Bu X, Chu C, Zhang J, Kolodziejczyk A, Fan Y, Chan NT, Ma L, Liu J, Wang D, Dai X, Liu H, Ono M, Nakanishi A, Inuzuka H, North BJ, Huang YH, Sharma S, Geng Y, Xu W, Liu XS, Li L, Miki Y, Sicinski P, Freeman GJ, Wei W. Acetylation-dependent regulation of PD-L1 nuclear translocation dictates the efficacy of anti-PD-1 immunotherapy. Nat Cell Biol. 2020 Sep;22(9):1064-1075. doi: 10.1038/s41556-020-0562-4. Epub 2020 Aug 24. PMID 32839551
- [Background] Salgia NJ, Bergerot PG, Maia MC, Dizman N, Hsu J, Gillece JD, Folkerts M, Reining L, Trent J, Highlander SK, Pal SK. Stool Microbiome Profiling of Patients with Metastatic Renal Cell Carcinoma Receiving Anti-PD-1 Immune Checkpoint Inhibitors. Eur Urol. 2020 Oct;78(4):498-502. doi: 10.1016/j.eururo.2020.07.011. Epub 2020 Aug 19. PMID 32828600
- [Background] Tumeh PC, Harview CL, Yearley JH, Shintaku IP, Taylor EJ, Robert L, Chmielowski B, Spasic M, Henry G, Ciobanu V, West AN, Carmona M, Kivork C, Seja E, Cherry G, Gutierrez AJ, Grogan TR, Mateus C, Tomasic G, Glaspy JA, Emerson RO, Robins H, Pierce RH, Elashoff DA, Robert C, Ribas A. PD-1 blockade induces responses by inhibiting adaptive immune resistance. Nature. 2014 Nov 27;515(7528):568-71. doi: 10.1038/nature13954. PMID 25428505